CLINICAL TRIAL: NCT06767124
Title: Simultaneous PET/MR Imaging of Brain Glucose and Oxygen Metabolism to Assess Energy Deficits Related to Alzheimer's Disease and the Response to Intervention
Brief Title: Supplementing Neuro-Energy to Aid Cognition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 126350; 1R01NS131235-01A1 (NIH)
Record Dates: First submitted 2025-01-06; First posted 2025-01-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease and Related Dementias (ADRD)
Keywords: PET/MR, Keytone Supplement, Brain Energy Metabolism
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Each patient receives a placebo and the active treatment on separate occasions undergoing the same imaging protocol.
Who Masked: Participant
Masking Description: Participants will not know if they have consumed the keytone ester supplement drink or a placebo drink.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alzheimer's Disease Patients - Treatment (Active Comparator): Patients within the Alzheimer's continuum will be selected based on the National Institute of Aging - Alzheimer's Association Diagnostic Framework and be either classified as having mild cognitive impairment or mild-to-moderate dementia. Participants will undergo two PET/MR sessions in which CMRGlu and CMRO2 will be imaged simultaneously by PET and qBOLD MRI. For validation, CMRO2 will also be imaged by PMROx prior to FDG injection. The study will follow a crossover design in which participants will receive ketogenic supplement prior to imaging.
  Interventions: Dietary Supplement: Ketogenic Supplement
- Alzheimer's Disease Patients - Placebo (Placebo Comparator): Patients within the Alzheimer's continuum will be selected based on the National Institute of Aging - Alzheimer's Association Diagnostic Framework and be either classified as having mild cognitive impairment or mild-to-moderate dementia. Participants will undergo two PET/MR sessions in which CMRGlu and CMRO2 will be imaged simultaneously by PET and qBOLD MRI. For validation, CMRO2 will also be imaged by PMROx prior to FDG injection. The study will follow a crossover design in which participants will receive a placebo drink prior to imaging.
  Interventions: Other: Placebo Drink

INTERVENTIONS:
Dietary Supplement: Ketogenic Supplement — Commercially available ketone ester drink
  Other Names: Ketone-IQTM
  Arms: Alzheimer's Disease Patients - Treatment
Other: Placebo Drink — Placebo drink containing sunflower oil.
  Arms: Alzheimer's Disease Patients - Placebo

SUMMARY:
It is projected that by 2030, one in every five Americans will be of retirement age, and this demographic shift is expected to result in more people suffering from dementia. A key feature of the brain is its need for a constant supply of glucose and oxygen to meet the high energy costs of mental activity. This study aims to develop clinically practical, noninvasive imaging methods based on combined positron emission tomography and magnetic resonance imaging to assess brain energy in order to better understand how this critical component of brain health is impacted by aging.

DETAILED DESCRIPTION:
There are now close to six million people in the Unites States living with dementia and this number is only expected to grow as the population continues to age. The current lack of effective treatments for Alzheimer's disease (AD) speaks to the need to better understand the multiple factors that contribute to this complex disease. There is growing evidence that age-related metabolic dysfunction in the brain plays a role in the disease's etiology. This concept has led to treatments aimed at improving brain energy production. Notably, ketogenic dietary supplements have been shown to increase brain ketone metabolism and improve cognitive performance in AD patients. However, the overall benefits to brain metabolism in the AD brain are unknown given the complexity of imaging both oxygen and glucose metabolism in a single session by positron emission tomography (PET). Taking advantage of hybrid PET/MR imaging, this study will combine PET and MRI methods to investigate the effects of a ketogenic supplement on brain oxygen and glucose metabolism in AD patients.

ELIGIBILITY:
Inclusion Criteria - Healthy Participants: Males and females, Age 21 - 80 years, BMI of 18.5-30

Inclusion Criteria - Alzheimer's Disease Participants: Positive amyloid and tau biomarkers (as noted by PET imaging, cerebrospinal fluid or blood), Mild cognitive impairment or mild-to-moderate dementia, BMI of 18.5-30

Exclusion Criteria: Contraindications to MRI (claustrophobia, metal implants, pacemakers, etc.), Pregnant or breastfeeding women, Neurological disease (healthy participants only), Mental illness, Overt cardio- or neurovascular disease, Recent participation in any procedure(s) involving radioactive agents

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral Metabolic Rate of Oxygen (CMRO2) | CMRO2 will be measured in both imaging sessions (placebo and ketosis)
  Statistical analysis of imaging data sets under placebo and ketosis conditions will be used to investigate increases in regional CMRO2 caused by ketosis.
Cerebral Metabolic Rate of Glucose (CMRGlu) | CMRGlu will be measued in both imaging session (placebo and ketosis)
  Statistical analysis of imaging data sets under palcebo and ketosis conditions will be used to investigate changes in regional CMRGlu caused by ketosis. Unlikek CMRO2, no difference in CMRGlu is expected between the two conditions for Alzheimer's patients.

SECONDARY OUTCOMES:
Cognitive Function | Baseline and 7 Days
  A psychometrist will assess baseline cognition using the Mini-Mental State Examination, the Montreal Cognitive Assessment, and the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog). The ADAS-cog will be repeated at the end of the second imaging session to test the potential cognitive benefits of the ketogenic supplement.

CONTACTS AND LOCATIONS:
Overall Officials: Keith St Lawrence, PhD, Principal Investigator — Lawson Research Institute
Locations (1):
- Lawson Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data sets to be shared include imaging data and participant demographics. Data will be made publicly available through the data sharing and archiving platform OpenNeuro.
Supporting Information: Study Protocol, SAP
Time Frame: Data release will follow a 36-month optional embargo to allow time for publication in a peer-reviewed journal.
Access Criteria: Data submitted to OpenNeuro are first associated with metadata from the BIDS dataset and with submitter-provided metadata, then indexed for searching. Copies of absorbed content -- from each submitted dataset version -- are subsequently assigned persistent digital object identifiers (DOIs).
  Datasets will be made publicly available through OpenNeuro with nominal restrictions using multiple open protocols. Prior to being made public, access to a dataset is controlled through strict authentication policies and an isolated storage backend to further guard against unintended access.